CLINICAL TRIAL: NCT04326036
Title: Use of cSVF For Residual Lung Damage (COPD/Fibrotic Lung Disease After Symptomatic COVID-19 Infection For Residual Pulmonary Injury or Post-Adult Respiratory Distress Syndrome Following Viral (SARS-Co-2) Infection
Brief Title: Use of cSVF Via IV Deployment for Residual Lung Damage After Symptomatic COVID-19 Infection
Acronym: GARM-COVID19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Black Tie Medical, Inc. (Industry)
Collaborators: Robert W. Alexander, MD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GARM COVID19
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Alveolar Proteinosis; COPD; Idiopathic Pulmonary Fibrosis; Viral Pneumonia; Coronavirus Infection; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis; Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Pneumonia, Viral; Coronavirus Infections; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Lipoaspiration (Experimental): Closed sterile, disposable microcannula of small volume adipose tissue, including the stromal vascular fraction (SVF) (cells and stromal tissue
  Interventions: Procedure: Microcannula Harvest Adipose Derived tissue stromal vascular fraction (tSVF)
- Isolation & Concentration of cSVF (Experimental): Isolation & Concentration of cellular stromal vascular fraction (cSVF) using Healeon Centricyte 1000 Centrifuge, incubator and shaker plate with sterile Liberase enzyme (Roche Medical) per manufacturer protocols
  Interventions: Device: Centricyte 1000; Drug: Liberase Enzyme (Roche)
- Delivery cSVF via Intravenous (Experimental): cSVF from Arm 2 is suspended in a 250 cc of sterile Normal Saline IV solution and deployed though 150 micron in-line filtration and intravenous route over 30-60 minute timeframe
  Interventions: Procedure: IV Deployment Of cSVF In Sterile Normal Saline IV Solution; Drug: Sterile Normal Saline for Intravenous Use
- Liberase TM (Other): Use of sterile Liberase TM enzyme to allow cSVF separation and isolation
  Interventions: Device: Centricyte 1000; Drug: Liberase Enzyme (Roche)
- Sterile Normal Saline (Other): 250 cc of sterile Normal Saline for Intravenous with sterile 150 micron in-line filtration for suspension of the concentrated cSVF and deployment IV
  Interventions: Procedure: IV Deployment Of cSVF In Sterile Normal Saline IV Solution; Drug: Sterile Normal Saline for Intravenous Use

INTERVENTIONS:
Procedure: Microcannula Harvest Adipose Derived tissue stromal vascular fraction (tSVF) — Use of Disposable Microcannula Closed System (Tulip Med, 2.2 mm) Harvest of Autologous Adipose Stroma and Stem/Stromal Cell Content
  Arms: Lipoaspiration
Device: Centricyte 1000 — Centricyte 1000 (Healeon Medical) Digestive (sterile Roche Liberase TM) Isolation/Concentration Protocol, Rinsing/Neutralization, and Pelletize the cSVF For Deployment Via Sterile Saline IV fluid Standard Protocol
  Arms: Isolation & Concentration of cSVF; Liberase TM
Procedure: IV Deployment Of cSVF In Sterile Normal Saline IV Solution — Sterile Normal Saline Suspension cSVF in 250cc for Intravenous Delivery Including Use of 150 micron in-line filtration
  Arms: Delivery cSVF via Intravenous; Sterile Normal Saline
Drug: Liberase Enzyme (Roche) — Sterile Collagenase Blend to separate cSVF from the AD-SVF
  Other Names: Proteolytic Emzyme
  Arms: Isolation & Concentration of cSVF; Liberase TM
Drug: Sterile Normal Saline for Intravenous Use — Sterile Normal Saline IV solution to provide suspension of cSVF in 250 cc via standard IV line, including sterile 150 micron in-line standard filter
  Other Names: Suspensory Fluid for cSVF
  Arms: Delivery cSVF via Intravenous; Sterile Normal Saline

SUMMARY:
COVID-19 Viral Global Pandemic resulting in post-infection pulmonary damage, including Fibrotic Lung Disease due to inflammatory and reactive protein secretions damaging pulmonary alveolar structure and functionality. A short review includes:

* Early December, 2019 - A pneumonia of unknown cause was detected in Wuhan, China, and was reported to the World Health Organization (WHO) Country Office.
* January 30th, 2020 - The outbreak was declared a Public Health Emergency of International Concern.
* February 7th, 2020 - 34-year-old Ophthalmologist who first identified a SARS-like coronavirus) dies from the same virus.
* February 11th, 2020 - WHO announces a name for the new coronavirus disease: COVID-19.
* February 19th, 2020 - The U.S. has its first outbreak in a Seattle nursing home which were complicated with loss of lives..
* March 11th, 2020 - WHO declares the virus a pandemic and in less than three months, from the time when this virus was first detected, the virus has spread across the entire planet with cases identified in every country including Greenland.
* March 21st, 2020 - Emerging Infectious Disease estimates the risk for death in Wuhan reached values as high as 12% in the epicenter of the epidemic and ≈1% in other, more mildly affected areas. The elevated death risk estimates are probably associated with a breakdown of the healthcare system, indicating that enhanced public health interventions, including social distancing and movement restrictions, should be implemented to bring the COVID-19 epidemic under control." March 21st 2020 -Much of the United States is currently under some form of self- or mandatory quarantine as testing abilities ramp up..

March 24th, 2020 - Hot spots are evolving and identified, particularly in the areas of New York-New Jersey, Washington, and California.

Immediate attention is turned to testing, diagnosis, epidemiological containment, clinical trials for drug testing started, and work on a long-term vaccine started.

The recovering patients are presenting with mild to severe lung impairment as a result of the viral attack on the alveolar and lung tissues. Clinically significant impairment of pulmonary function appears to be a permanent finding as a direct result of the interstitial lung damage and inflammatory changes that accompanied.

This Phase 0, first-in-kind for humans, is use of autologous, cellular stromal vascular fraction (cSVF) deployed intravenously to examine the anti-inflammatory and structural potential to improve the residual, permanent damaged alveolar tissues of the lungs.

DETAILED DESCRIPTION:
COVID-19 Viral Global Pandemic resulting in post-infection pulmonary damage, including Fibrotic Lung Disease due to inflammatory and reactive protein secretions damaging pulmonary alveolar structure and functionality. A short review includes:

* Early December, 2019 - A pneumonia of unknown cause was detected in Wuhan, China, and was reported to the World Health Organization (WHO) Country Office.
* January 30th, 2020 - The outbreak was declared a Public Health Emergency of International Concern.
* February 7th, 2020 - 34-year-old Ophthalmologist who first identified a SARS-like coronavirus) dies from the same virus.
* February 11th, 2020 - WHO announces a name for the new coronavirus disease: COVID-19.
* February 19th, 2020 - The U.S. has its first outbreak in a Seattle nursing home which were complicated with loss of lives..
* March 11th, 2020 - WHO declares the virus a pandemic and in less than three months, from the time when this virus was first detected, the virus has spread across the entire planet with cases identified in every country including Greenland.
* March 11th, 2020 - As of this date, Over 60% of all COVID-19 deaths in the U.S. can be traced to that single nursing home in Seattle.
* March 11th, 2020 - Dr. Fauci from the National Institutes of Health (NIH) states, "If you count all the estimated cases of people who may have it but haven't been diagnosed yet, the mortality rate is probably closer to 1%," he said, "which means it's 10 times more lethal than the seasonal flu."
* March 21st, 2020 - The U.S. has 24,105 active cases, 301 deaths, and 171 patients declared recovered, a number which has since massively increased within the United States and Globally.
* March 21st, 2020 - Emerging Infectious Disease estimates the risk for death in Wuhan reached values as high as 12% in the epicenter of the epidemic and ≈1% in other, more mildly affected areas. The elevated death risk estimates are probably associated with a breakdown of the healthcare system, indicating that enhanced public health interventions, including social distancing and movement restrictions, should be implemented to bring the COVID-19 epidemic under control." March 21st 2020 -Much of the United States is currently under some form of self- or mandatory quarantine as testing abilities ramp up..

March 24th, 2020 - Hot spots are evolving and identified, particularly in the areas of New York-New Jersey, Washington, and California

Immediate attention is turned to testing, diagnosis, epidemiological containment, clinical trials for drug testing started, and work on a long-term vaccine started.

The recovering patients are presenting with mild to severe lung impairment as a result of the viral attack on the alveolar and lung tissues. Clinically significant impairment of pulmonary function appears to be a permanent finding as a direct result of the interstitial lung damage and inflammatory changes that accompanied.

This Phase 0, first-in-kind for humans, is use of autologous, cSVF deployed intravenously to examine the anti-inflammatory and structural potential to improve the residual damaged tissues.

Previous utilization of cSVF remains in Clinical Trials at this moment for uses in Chronic Obstructive Pulmonary Disease (COPD) and Idiopathic Pulmonary Fibrotic Lung disorders, showing encouraging safety profile and clinical efficacy. It is the intention of this study, driven by the ongoing pandemic as a direct causative etiology for permanent lung damage within the oxygen/carbon dioxide exchange resulting the the direct alveolar disruption and scarring reaction.

The inflammatory mediation, autoimmune modulatory capabilities, and revascularization potentials of the cSVF is becoming well recognized and documented in peer-reviewed literature and in scientific studies.

Due to the urgency presented from the ongoing CoronaVirus pandemic, many patients that survive experience demonstrate direct pulmonary damage residua. There is available a relative new technology offered by Fluidda Inc in European Union (EU) known as "Functional Respiratory Imaging (FRI) and examines pulmonary function and vascular capabilities in damaged lung tissues. This study examines the lung baseline (post-infection), and at 3 and 6 month intervals post-cSVF treatment to examine the functional airway configuration and efficiency at those intervals.

Sporadic reports of use of stem cells or stem/stromal cells have revealed some positive clinical outcomes, although not within a traditional randomized trial format at this point in time. This study proposed in the specific situation of permanent residual dysfunction created by the SARS-Co2 (Coronavirus) infection is felt to warrant a pilot study using the cSVF that is in current Clinical Trials, which, at this point presents a very good safety profile with the absence of adverse event (AE) or severe adverse events (SAE) as yet reported by the trials.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed and documented Coronaviral (COVID-19) infection history with involvement of lung tissues
* Must be clear of any viral shed residual confirmed by negative viral testing protocol accepted by the Center for Disease Control (CDC) and/or the FDA
* Must have discharge confirmation from infectious disease managing Provider declaring freedom of viral load or active infection
* Must have a written Medical History of Physical and discharge summary (if hospitalized) from appropriate Center or Licensed Medical Provider
* Must agree to provide a HRCT LUNG study done at baseline (before), 3 months and 6 months
* Must be able to provide full Informed Consent (ICF)

Exclusion Criteria:

* Active or positive testing of COVID-19 With Clinical Report and Discharge Summary from Hospital or Treatment Facility
* Lung disorder without prior confirmation by approved test protocol of history of COVID-19
* Patient health or condition deemed dangerous or inappropriate for transport, exceeding acceptable stress for transport or care needed to achieve access to the clinical facility, at the discretion of the Providers
* Expected lifespan of < 6 months
* Serious of life threatening co-morbidities, that in the opinion of the investigators, may compromise the safety or compliance with the study guidelines and tracking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 month
  Reporting of Adverse Events or Severe Adverse Events Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Pulmonary Function Analysis | baseline, 3 Month, 6 months
  High Resolution Computerized Tomography of Lung (HRCT Lung) for Fluidda Analysis comparative at baseline and 3 and 6 months post-treatment comparative analytics
Digital Oximetry | 3 months, 6 months
  Finger Pulse Oximetry taken before and after 6 minute walk on level ground, compare desaturation tendency

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Alexander, MD, Study Chair — Global Alliance Regenerative Medicine
Locations (1):
- Robert W. Alexander, MD, FICS, LLC, Stevensville, Montana, United States

IPD SHARING:
Plan to Share IPD: No
In discussion phase

REFERENCES:
- [Background] Alexander, Robert W., Overview of Cellular Stromal Vascular Fraction (cSVF) & Biocellular Uses of Stem/Stromal Cells & Matrix (tSVF + HD-PRP) in Regenerative Medicine, Aesthetic Medicine and Plastic Surgery. 2019, S1003, DOI: 10.24966/SRDT-2060/S1003.
- [Background] Alexander, Robert W., Understanding Adipose-Derived Stromal Vascular Fraction (AD-SVF) Cell Biology and Use on the Basis of Cellular, Chemical, Structural and Paracrine Components. (2012), J of Prolotherapy, 4: 855-869.
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Li G, De Clercq E. Therapeutic options for the 2019 novel coronavirus (2019-nCoV). Nat Rev Drug Discov. 2020 Mar;19(3):149-150. doi: 10.1038/d41573-020-00016-0. No abstract available. PMID 32127666
- [Background] Wu K, Peng G, Wilken M, Geraghty RJ, Li F. Mechanisms of host receptor adaptation by severe acute respiratory syndrome coronavirus. J Biol Chem. 2012 Mar 16;287(12):8904-11. doi: 10.1074/jbc.M111.325803. Epub 2012 Jan 30. PMID 22291007
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Ding Y, He L, Zhang Q, Huang Z, Che X, Hou J, Wang H, Shen H, Qiu L, Li Z, Geng J, Cai J, Han H, Li X, Kang W, Weng D, Liang P, Jiang S. Organ distribution of severe acute respiratory syndrome (SARS) associated coronavirus (SARS-CoV) in SARS patients: implications for pathogenesis and virus transmission pathways. J Pathol. 2004 Jun;203(2):622-30. doi: 10.1002/path.1560. PMID 15141376
- [Background] Kawase M, Shirato K, van der Hoek L, Taguchi F, Matsuyama S. Simultaneous treatment of human bronchial epithelial cells with serine and cysteine protease inhibitors prevents severe acute respiratory syndrome coronavirus entry. J Virol. 2012 Jun;86(12):6537-45. doi: 10.1128/JVI.00094-12. Epub 2012 Apr 11. PMID 22496216
- [Background] Zhang R, Pan Y, Fanelli V, Wu S, Luo AA, Islam D, Han B, Mao P, Ghazarian M, Zeng W, Spieth PM, Wang D, Khang J, Mo H, Liu X, Uhlig S, Liu M, Laffey J, Slutsky AS, Li Y, Zhang H. Mechanical Stress and the Induction of Lung Fibrosis via the Midkine Signaling Pathway. Am J Respir Crit Care Med. 2015 Aug 1;192(3):315-23. doi: 10.1164/rccm.201412-2326OC. PMID 25945397